CLINICAL TRIAL: NCT02888782
Title: Optimizing Medication Therapy Outcomes for Complex Patients Transitioning From Acute to Primary Care
Brief Title: Optimizing Medication Therapy for Patients Recently Discharged From Hospital
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Program Restructured
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Deborah Kelly, Associate Professor and Special Advisor of Innovation, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HREB-2016.221
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacist Consultation (Experimental): Meet with pharmacist for consultation in addition to regular physician follow up
  Interventions: Other: Pharmacist Consultation
- Control (No Intervention): Receive regular physician follow up

INTERVENTIONS:
Other: Pharmacist Consultation
  Arms: Pharmacist Consultation

SUMMARY:
Patients who are discharged from hospital can be overwhelmed when they suddenly have to manage new conditions or medications. These changes can be particularly difficult for people on many medications or with multiple health conditions. There is a real risk that this will lead to emergency room visits, hospital readmission, and even death. In addition to endangering patients, these adverse events are very costly to the healthcare system. The good news is that these events can be preventable if patients receive care that is better coordinated.

Patient-oriented research will be conducted to determine if a pharmacist-led medication therapy management service can improve health outcomes of 'medically complex' patients transitioning from acute to primary care in Newfoundland and Labrador (NL). This a more comprehensive service than their community pharmacist would normally provide. The program will use a new Pharmacist Clinic service to provide care and support which does not currently exist for patients in NL after they leave hospital. After discharge, patients will be randomly divided into two groups: one group will receive care as usual from their doctor; the other group will have their medications assessed by a clinic pharmacist within one week of hospital discharge along with their usual care from their doctor. The two groups will be compared to determine whether specialized pharmacist services after hospital discharge is satisfactory to patients/providers, improves patient health, and reduces emergency room visits, hospital readmissions, and repeat trips to the doctor. If successful, this project will help ensure that patients are taking the right medications in the right way, improving individual health and making better use of healthcare system resources.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of age or older
2. Admitted to a General Medicine ward
3. Take 5 or more chronic medications

Exclusion Criteria:

1. Discharge to a long term care facility
2. Life expectancy less than 3 months
3. Have entered palliative care
4. Cognitive impairment (unless a responsible caregiver can provide consent and assist in participation)
5. Non-English speaking
6. Unable to provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Composite Hospital Utilization Rate | 30 days post discharge
  A composite score of hospital readmission rate and ER visits

SECONDARY OUTCOMES:
Number of Emergency Room Visits | 30 days post discharge
Number of Emergency Room Visits | 60 days post discharge
Number of Emergency Room Visits | 90 days post discharge
Rehospitalization Rate | 30 days post discharge
Rehospitalization Rate | 60 days post discharge
Rehospitalization Rate | 90 days post discharge
Mortality Rate | 30 days post discharge
Mortality Rate | 60 days post discharge
Mortality Rate | 90 days post discharge
Frequency of Family Physician Visits | 30 days post discharge
Frequency of Family Physician Visits | 60 days post discharge
Frequency of Family Physician Visits | 90 days post discharge

OTHER OUTCOMES:
Patient Satisfaction Survey | Collected 3 - 6 months after study enrollment
  Measured using a Likert scale questionnaire
Pharmacist Satisfaction Survey | Collected at the end of study period (12-15 months)
  Measured using a Likert scale questionnaire
Physician Satisfaction Survey | Collected at the end of study period (12-15 months)
  Measured using a Likert scale questionnaire
Patient quality of life Short Form Health Survey | Collected at time of hospital discharge
  Measured using a Short Form Health Survey (SF-36)
Patient quality of life Short Form Health Survey | Collected at 30, 60 and 90 days post hospital discharge
  Measured using a Short Form Health Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Kelly, PharmD, Principal Investigator — Memorial Univeristy of Newfoundland
Locations (2):
- Canada (2):
  - Health Sciences Center, St. John's, Newfoundland and Labrador
  - St. Clares Mercy Hospital, St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: No